CLINICAL TRIAL: NCT01637675
Title: Clinical Study of Effects of Sodium Tanshinone IIA Sulfonate on Pulmonary Hypertension
Brief Title: Efficacy and Safety Study of Sodium Tanshinone IIA Sulfonate on Pulmonary Hypertension
Acronym: STS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Jiangsu Carefree Pharmaceutical Co., Ltd. (Industry); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Guangdong Provincial People's Hospital (Other); Sir Run Run Shaw Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Dongguan People's Hospital (Other Government); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Beijing Chao Yang Hospital (Other); Beijing Anzhen Hospital (Other); The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Nanshan Zhong, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STS-PH01
Record Dates: First submitted 2012-07-01; First posted 2012-07-11 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension; Cardiovascular Diseases; Lung Diseases; Tanshinone IIA Sulfonate
Keywords: sodium tanshinone IIA sulfonate; pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Cardiovascular Diseases; Lung Diseases | interventions — Sildenafil Citrate; tanshinone II A sodium sulfonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20 mg sildenafil citrate tablets by mouth (Active Comparator): 20 mg sildenafil citrate tablets by mouth three times a day for 8 weeks
  Interventions: Drug: 20 mg sildenafil citrate by mouth
- sodium tanshinone IIA sulfonate, sildenafil citrate tablets (Experimental): sodium Tanshinone IIA sulfonate injection 80 mg diluted with 5% glucose solution(0.9% sodium chloride injection also permitted if necessary) 250ml ivdrip once a day for 8 weeks,20mg sildenafil citrate tablets by mouth three times a day for the same duration
  Interventions: Drug: sodium tanshinone IIA sulfonate diluted with 5% glucose solution,20mg sildenafil citrate by mouth

INTERVENTIONS:
Drug: 20 mg sildenafil citrate by mouth — 20 mg sildenafil citrate tablets by mouth three times a day for 8 weeks
  Other Names: Viagra
  Arms: 20 mg sildenafil citrate tablets by mouth
Drug: sodium tanshinone IIA sulfonate diluted with 5% glucose solution,20mg sildenafil citrate by mouth — sodium Tanshinone IIA sulfonate injection 80 mg diluted with 5% glucose solution(0.9% sodium chloride injection will also be permitted if necessary) 250ml iv drip once a day for 8 weeks,as well as 20mg sildenafil citrate tablets by mouth three times a day for the same duration of treatment
  Other Names: Sodium tanshinone IIA sulfonate injection; Viagra
  Arms: sodium tanshinone IIA sulfonate, sildenafil citrate tablets

SUMMARY:
Sodium tanshinone IIA sulfonate (STS) is a water-soluble derivative of tanshinone IIA isolated as the main pharmacologically active natural compound from a traditional Chinese herbal medicine,the dried root of Salvia miltiorrhiza Bunge known as Danshen. Danshen has been known for the function of improving body functions such as activating blood circulation and removing blood stasis according to the theory of traditional Chinese medicine. Danshen and its various formula products including STS have been long-time widely used in oriental countries, especially China to treat various inflammatory and cardiovascular diseases for its pharmacological actions, including vasodilatation, anticoagulation, anti-inflammation, and free radical scavenging,with negligible adverse effects observed.

The investigator's objective is to evaluate whether STS exhibits beneficial effects on pulmonary hypertension. This is a randomized, controlled, multicentre clinical trial study. 90 patients with pulmonary hypertension will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the condition of mean pulmonary arterial pressure (mPAP) ≥25 mmHg at seal level at rest and pulmonary capillary wedge pressure(PCWP)≤15mmHg;
2. Category 1 or 4 of PH in stable stage according to 2008 Dana Point Conference,including the idiopathic, hereditary, drugs and toxins induced, associated with connective tissue disease or congenital heart disease, and chronic thromboembolic pulmonary arterial hypertension(PAH) ;
3. Male or female between 15 to 70 years old;
4. WHO pulmonary hypertension functional class II or III;
5. The baseline 6-minute walk distance between 150-550 m;
6. Patients' condition should be stable for more than one month after basic treatment; For those patients with congenital heart disease, surgery should have been performed six months or more before they are enrolled in the study;
7. Patients receiving sildenafil treatment only previously, or those without target drugs treatment during the past 3 months;
8. Patients or their guardians should agree with this clinical trail and medical informed consent of the trial should be signed.

Exclusion Criteria:

1. Unavailable or limited legal capacity;
2. Pregnant or lactational women;
3. Important organs with severe diseases;
4. Mental or physical disability;
5. With suspected or indeed alcohol, drug abuse history;
6. With allergic constitution, with two or more drugs or foods allergy history or those who are allergic to any components of the experimental drugs;
7. With both aspartate aminotransferase (AST) and glutamic-pyruvic transaminase (ALT) more than three times of the upper limit of normal in liver function test and Ccr≤50ml/min in kidney function test;
8. Those with systemic blood pressure<90/50 mmHg, or those uncontrolled dangerous hypertension(BP>170/110 mmHg);
9. Patients at active stages of infectious or other diseases such as hepatitis A, hepatitis B, AIDS, tuberculosis, and some connective tissue diseases;
10. Patients with severe infection, especially pulmonary infection;
11. Patients with shock or astable hemodynamics with other causes;
12. Patients with hepatic cirrhosis, and hepatic cirrhosis induced portal hypertension;
13. Patients with severe hemorrhage, and hemorrhagic tendency;
14. Patients who need to take or be taking drugs possible or indeed affecting this trial;
15. Patients cannot accomplish required items (especially 6MWD) because of acute/chronic organic disease (excluding dyspnea) or other illnesses such as lower extremity diseases;
16. Patients with any other conditions considered cannot be recruited.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
mPAP by right heart catheterization | At the end of 0- and 8-week trial
  To assess if sodium Tanshinone IIA sulfonate decreases mean pulmonary arterial pressure.

SECONDARY OUTCOMES:
WHO functional class of pulmonary hypertension(PH) | At the end of 0-,2-, 4-,6- and 8-week of trial
Borg dyspnea score | At the end of 0-, 2-,4-,6- and 8-week trial
Minnesota living with heart failure questionnaire | At the end of 0-,2-, 4-,6- and 8-week trial
6-minute walk distance (6MWD) | At the end of 0-, 2-, 4-, 6- and 8-week trial
  To assess if sodium Tanshinone IIA sulfonate improves the exercise capacity of patients with pulmonary hypertension.
Pulmonary vascular resistance(PVR) measured by right heart catheterization | At the end of 0- and 8-week trial
  PVR is used to evaluate whether STS decreases mPAP or increases pulmonary circulatory blood flow.

OTHER OUTCOMES:
The level of N terminal-proBNP(NT-proBNP),cardiac troponin I(cTnI) and uric acid(UA) in serum | At the end of 0-,4- and 8-week trial
  The three indicators are used to evaluate whether STS alleviates right heart failure.
Indicators monitoring STS safety | At the end of 0-,4- and 8-week trial
  The blood routine test,urine routine test,liver and kidney function and blood clotting function will be examined and some worsening events,such as death,PH aggravation,need to add other unscheduled target drugs,need to be hospitalized or prolonged hospitalization,lung and/or heart transplantation and/or any other severe adverse events surely or very likely due to STS,will be closely observed as the safety indications of STS.
Other hemodynamic parameters measured by right heart catheterization | At the end of 0- and 8-week trial
  To evaluate whether STS has beneficial effects on hemodynamic parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] He X, Yang F, Wu Y, Lu J, Gao X, Zhu X, Yang J, Liu S, Xiao G, Pan X. Identification of tanshinone I as cap-dependent endonuclease inhibitor with broad-spectrum antiviral effect. J Virol. 2023 Oct 31;97(10):e0079623. doi: 10.1128/jvi.00796-23. Epub 2023 Sep 21. PMID 37732786